CLINICAL TRIAL: NCT00485420
Title: Using the Internet to Provide Disease Management and Improve Compliance Among Bipolar and Depressed Patients
Brief Title: eCare for Moods: An Internet-based Management Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CN-02EHunk-02-H
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Internet based disease management program
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator): Member with recurrent or chronic depression receives usual specialty mental health care
  Interventions: Other: Internet based disease management program
- Internet-based disease managment program (Experimental): Usual care is augmented with internet based education, self monitoring and clinical monitoring
  Interventions: Other: Internet based disease management program

INTERVENTIONS:
Other: Internet based disease management program — Usual Care is augmented with internet-based education, self-monitoring and clinician monitoring
  Other Names: Care management via the internet

SUMMARY:
The study aim is to explore the effect of a comprehensive Internet-based disease management program for bipolar disorder and recurrent or chronic major depression on clinical outcomes and satisfaction with care.

DETAILED DESCRIPTION:
This study is a randomized controlled trial that includes 404 subjects, 300 subjects with bipolar disorder and 104 subjects with recurrent or chronic major depressive disorder. The study subject diagnostic groups (bipolar and depressive) are separately randomized to either usual care or to eCare and the data collected from the two diagnostic groups are analyzed separately.

All subjects randomized to the eCare intervention are assigned an eCare nurse care manager in addition to one year of access to an Internet-delivered care management and patient self-management program. While both diagnostic groups receive similar Internet-delivered services for depression, the subjects with bipolar disorder receive special services for bipolar disorder. All subjects randomized to usual care will receive their normal psychiatric care and do not have access to the website.

Study subjects are followed for 24 months and outcome measurements are taken every six months by telephone interviewers blinded to treatment assignment. Specific measures include depression and mania symptoms, severity, adherence with medication, general health, functioning at work and at home, satisfaction with care, and confidence in coping with their disorder. The primary outcomes for patients with bipolar disorder are the severity of depression and the severity of mania over time. The primary outcome for patients with recurrent or chronic depression is the severity of depression over time. The hypothesis is that Internet-based care management will have a favorable effect on the burden of bipolar disorder and/or on recurrent/chronic depression over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar or recurrent major depressive disorder and access to a computer

Exclusion Criteria:

* No diagnosis of bipolar or recurrent major depressive disorder, no computer access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2002-09; Primary Completion 2009-09 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Reduction of severity of mania and depression symptoms and reduction in frequency of occurrence depression symptoms | Two years

SECONDARY OUTCOMES:
Satisfaction with medical care | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Enid M Hunkeler, MA, Principal Investigator — Kaiser Permanente Division of Research